CLINICAL TRIAL: NCT01632527
Title: Phase I/II Study of the Safety and Preliminary Efficacy of Human Central Nervous System Stem Cells (HuCNS-SC) Subretinal Transplantation in Subjects With Geographic Atrophy of Age-Related Macular Degeneration
Brief Title: Study of Human Central Nervous System Stem Cells (HuCNS-SC) in Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StemCells CL-N01-AMD
Record Dates: First submitted 2012-06-21; First posted 2012-07-03 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Age Related Macular Degeneration; Macular Degeneration; AMD
Keywords: Age-Related Macular Degeneration; Dry AMD with GA; Geographic Atrophy of Age-Related Macular Degeneration; Stem Cell Transplantation; Stem Cell transplant; Stem cells for AMD; Human neural stem cells; multipotent stem cells; Macular Degeneration; Dry AMD; Human central nervous system stemcells; dry age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HuCNS-SC (Experimental): HuCNS-SC cells
  Interventions: Drug: HuCNS-SC cells

INTERVENTIONS:
Drug: HuCNS-SC cells — HuCNS-SC cells transplantation directly into the subretinal space of one eye (Study eye) in a single transplant procedure.
  Other Names: Human Central Nervous System Stem Cells

SUMMARY:
The purpose of this Phase I/II study is to investigate the safety and preliminary efficacy of unilateral subretinal transplantation of HuCNS-SC cells in subjects with geographic atrophy secondary to age-related macular degeneration.

DETAILED DESCRIPTION:
This study is an open-label dose-escalation investigation of the safety and preliminary efficacy of unilateral subretinal transplantation of HuCNS-SC cells in subjects with Geographic Atrophy secondary to Age-Related Macular Degeneration (AMD). Subjects will be enrolled based on specific inclusion/exclusion criteria and evaluated at regular post transplant intervals. The investigation will be divided into two sequential cohorts. Subjects will be enrolled into each cohort based on best-corrected visual acuity (BCVA) visual acuity as determined by the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) acuity test. BCVA of less than or equal to 20/400 in the Study Eye will be enrolled in Cohort I. Subjects with BCVA of 20/320 to 20/100 in the Study Eye will be enrolled in Cohort II. Cohort I will consist of four subjects who will undergo transplant with 200,000 cells followed by four subjects who will undergo transplant with 1 million cells. Cohort II will consist of 7 subjects who will undergo transplant with 1 million cells. An independent Data Monitoring Committee (DMC) will review accruing safety data for all subjects.

HuCNS-SC cells will be transplanted by a board-certified vitreoretinal surgeon. The transplantation will be conducted in the eye with the inferior best-corrected visual acuity (BCVA) (i.e., the Study Eye). Only the Study Eye will undergo transplantation. The HuCNS-SC cells will be administered into the subretinal space through a standard surgical approach.

Immunosuppressive agents will be administered orally to all subjects for a period of three months after surgery.

Subjects will be monitored frequently for a total of one year after HuCNS-SC cell transplantation. An additional four years of monitoring will be conducted in a separate follow-up study that will commence with the termination visit of the Phase I/II investigation. The follow-up study will be conducted as a separate investigation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of age-related macular degeneration with geographic atrophy (GA)
* Only patients with a specific degree and extent of GA will be eligible
* Subjects with best-corrected visual acuity (BCVA) of less than or equal to 20/400 in the Study Eye will be enrolled in Cohort I. Subjects with BCVA of 20/320 to 20/100 in the Study Eye will be enrolled in Cohort II
* No prior or current choroidal neovascularization in either eye
* Must have adequate care-giver support and access to medical care in the local community
* Able to provide written informed consent prior to any study related procedures
* Agree to comply in good faith with all conditions of the study and to attend all required study visits

Exclusion Criteria:

* Prior vitreal or retinal surgery
* Glaucoma
* Atrophic macular disease of any other cause
* Diabetic retinopathy or diabetic macular edema in either eye
* Previous organ, tissue or bone marrow transplantation
* Previous participation in a gene transfer or a cell transplant trial
* Autoimmune disease
* Allergy to tacrolimus, mycophenolate mofetil (MMF), scopolamine, Cyclogyl, Moxifloxacin, or Gatifloxacin
* Current or prior malignancy (or is on chemotherapy)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | One year following transplant surgery
  Descriptive analysis of frequency and types of adverse events experienced by each subject during the study period.

SECONDARY OUTCOMES:
Assessment of visual function changes from baseline | At frequent intervals for one year following transplantation
  Assessments will include BCVA by the E-ETDRS acuity test, fluorescein angiography and fundus photography, spectral domain ocular coherence tomography (OCT), microperimetry, multifocal electroretinography, contrast sensitivity, and a standardized questionnaire of visual function.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, M.D., Study Director — StemCells, Inc.
Locations (5):
- United States (5):
  - Retina-Vitreaous Associates Medical Group, Los Angeles, California
  - Byers Eye Institute at Stanford, Stanford Hospital and Clinics, Palo Alto, California
  - New York Eye and Ear Infirmary, New York, New York
  - Retina Research Institute of Texas, Abilene, Texas
  - Retina Foundation of the Southwest, Dallas, Texas

REFERENCES:
- See also: AMD and Retinal Disorders — http://www.stemcellsinc.com/Therapeutic-Programs/AMD-and-Retinal-Disorders.htm